CLINICAL TRIAL: NCT06868472
Title: Early Recovery After Surgery (ERAS)/Prehabilitation - Randomized Controlled Trial on the Implementation of ERAS/prehabilitation in Elective Reconstructive Shoulder Surgery
Acronym: Prehab
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Arasch Wafaisade (Other)
Responsible Party: Sponsor-Investigator, Prof. Arasch Wafaisade, Prof. Dr. med., University of Witten/Herdecke
Organization: University of Witten/Herdecke (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ethics number: 150/2024
Record Dates: First submitted 2025-02-07; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff
Keywords: Preoperative Exercise; Enhanced Recovery After Surgery
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehabilitation-Group (Active Comparator)
  Interventions: Procedure: Prehabilitation
- Control-Group (Placebo Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Prehabilitation — The waiting time until the operation is about 6 weeks. The intervention is carried out during this time:
  The intervention group receives a brochure with an evidence-based exercise program for the shoulder and shoulder girdle. The brochure contains pages in which the patient documents how the exercises are carried out. The exercise program is supplemented by information in the form of a video/Power Point presentation on: Anatomy/function, pain management, hospitalization and subsequent rehabilitation.
  After 2 and after 4 weeks, the physiotherapist who has explained the exercise program will contact you by telephone/zoom.
  Arms: Prehabilitation-Group
Procedure: Control — The control group receives a leaflet with general information for the period up to the operation (e.g. buy water-resistant plasters, arrange post-op physiotherapy appointments).
  Arms: Control-Group

SUMMARY:
The aim of this randomized controlled trial is to investigate whether the intervention can improve the clinical outcome and patient satisfaction in elective reconstructive shoulder surgeries. The study participants are adults with a diagnosed rotator cuff tear for which surgical treatment is planned. This main question is to be answered by the study:

• Does prehabilitation before elective shoulder surgeries lead to an improvement in postoperative outcomes and patient satisfaction compared to the control group?

The control group receives standard information about the hospital stay, while the intervention group undergoes the prehabilitation program in the approximately 6 weeks prior to surgery. This program includes:

* Information on the condition and pain management
* Recommendations for behavior modification
* A home exercise program Primary endpoint is the Western Ontario Rotator Cuff Index (WORC). The assessments are conducted at four time points: at study enrollment, immediately before surgery, and at 6, 12, and 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a traumatic or degenerative rupture of the rotator cuff with whom surgical treatment has been discussed in the shoulder clinic.

Exclusion Criteria:

* Pre-existing fracture of the upper arm or shoulder girdle, rheumatic arthritis/fibromyalgia, additional findings in the shoulder joint (instability, frozen shoulder), neurological disease, cognitive or speech impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-18 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | Inclusion in the study (T0), before surgery (T1); 6 months (T2), 12 months (T3) and 24 months (T4) after surgery
  The WORC Index is a self-administered questionnaire designed to assess the quality of life in individuals with rotator cuff tendinopathy. It consists of 21 items across five domains: Physical Symptoms, Sports and Recreation, Work, Lifestyle, and Emotions. Each item is rated on a visual analogue scale (VAS) from 0 to 100. The total score ranges from 0 to 2100, which can be converted to a percentage for easier interpretation. A higher percentage indicates better shoulder function. The WORC Index is widely used in clinical settings to evaluate symptoms, functional limitations, and treatment outcomes.

SECONDARY OUTCOMES:
Patient survey on Treatment satisfaction and willingness to recommend | before surgery (T1); 6 months (T2), 12 months (T3) and 24 months (T4) after surgery
  A brief, self-designed questionnaire was developed to measure overall satisfaction through patient satisfaction and willingness to recommend. It utilizes a 6-point Likert scale for responses.
EQ-5D quality of life questionnaire | Inclusion in the study (T0), before surgery (T1); 6 months (T2), 12 months (T3) and 24 months (T4) after surgery
  The EQ-5D is a standardized questionnaire developed by the EuroQol Research Foundation to measure health-related quality of life. It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each rated on a scale of severity. Additionally, it includes a visual analogue scale (EQ VAS) for the patient's self-rated health. The EQ-5D is widely used in clinical studies, health economics, and routine care to assess and compare quality of life across different health conditions and populations. It provides a simple, reliable, and internationally recognized tool for evaluating overall health status.
Constant Murely score for self-evaluation | Inclusion in the study (T0), before surgery (T1); 6 months (T2), 12 months (T3) and 24 months (T4) after surgery
  The Constant-Murley Score for self-evaluation, adapted by Boehm et al. in 2003, is a modified version of the original Constant-Murley Score that allows patients to independently assess their shoulder function. It includes parameters such as pain, activities of daily living, range of motion, and strength, scored on a standardized scale. This self-assessment tool provides a reliable and practical method for patients to evaluate their shoulder condition, enabling its use in clinical research and routine monitoring of treatment outcomes.
Subjective shoulder value | Inclusion in the study (T0), before surgery (T1); 6 months (T2), 12 months (T3) and 24 months (T4) after surgery
  The Subjective Shoulder Value (SSV) is a patient-reported numeric scale that reflects the subjective assessment of shoulder function. Patients rate their current shoulder function as a percentage compared to a normal, healthy shoulder, with 0% representing no function and 100% representing full, unrestricted function. Developed by Gilbart and Gerber in 2007, the SSV is a simple, quick, and reliable tool for evaluating subjective shoulder functionality. It is widely used in clinical studies and daily practice to monitor progress and document outcomes in shoulder conditions.
Survey on the use of painkillers | Inclusion in the study (T0), before surgery (T1); 6 months (T2), 12 months (T3) and 24 months (T4) after surgery
Survey on return to pre-operative sport | 6 months (T2), 12 months (T3) and 24 months (T4) after surgery
  Patients are asked whether they have resumed the sport they practiced before the operation and at what level of performance they have returned (same level, slightly reduced, significantly reduced or no sport). In addition, it is recorded whether the sport is an overhead sport.
Survey on return to preoperative occupation or daily responsibilities | 6 months (T2), 12 months (T3) and 24 months (T4) after surgery
  Patients are asked whether they have returned to their preoperative occupation or daily responsibilities. Additionally, it is recorded whether their work involves a desk job."
Examination for the presence of a re-rupture | 6 months (T2), 12 months (T3) and 24 months (T4) after surgery
  It is recorded whether a re-rupture has occurred postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken der Stadt Köln gGmbH, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No